CLINICAL TRIAL: NCT00299364
Title: Multi-Center, Randomized, Double-Blind, Parallel-Controlled Study on the Efficacy and Tolerability of Black Cohosh Vs Tibolone in Patients With Menopausal Symptoms
Brief Title: Comparison of the Efficacy and Tolerability of Black Cohosh Vs Tibolone in Patients With Menopausal Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Schaper & Bruemmer GmbH & Co KG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB-FEM0401
Record Dates: First submitted 2006-03-01; First posted 2006-03-06 (Estimated); Last update posted 2006-03-06 (Estimated); Status verified 2006-03

CONDITIONS: Menopause
Keywords: Climacteric symptoms; Black Cohosh; Efficacy; Safety
MeSH Terms: interventions — black cohosh root extract; tibolone

INTERVENTIONS:
Drug: Black Cohosh (iCR) or tibolone

SUMMARY:
The benefit-risk-balance of the isopropanolic Cimicifuga racemosa extract (iCR) is compared with tibolone in menopausal symptoms treatment. Menopausal patients aged 40 - 60 years and with a Kupperman Menopause Index (KMI) equal or more than 15 participate and were assigned to either iCR corresponding to 40 mg crude drug/day (n=122) or tibolone 2,5 mg/day (n=122) orally. The primary endpoint is the benefit-risk balance at end of treatment.

DETAILED DESCRIPTION:
The benefit-risk-balance of the isopropanolic Cimicifuga racemosa extract (iCR) is compared with tibolone in menopausal symptoms treatment. The randomized, double-blind, controlled 3-month study in 5 centres of 3 cities in China enrolled 244 menopausal patients aged 40 - 60 years and with a Kupperman Menopause Index (KMI) equal or more than 15. The participants were assigned to either iCR corresponding to 40 mg crude drug/day (n=122) or tibolone 2,5 mg/day (n=122) orally. The primary endpoint is the combination of the Mann-Whitney values (MWV) of the KMI and the frequency of adverse events (benefit-risk balance) at end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* between 40 years and 60 years of age
* spontaneous amenorrheic interval at least 5 months since the last regular menstruation
* for those patients with amenorrheic interval less than 12 months, the baseline level of E2 should not exceed 30 pg/ml
* Kupperman Menopause Index at least 15
* written informed consent
* good general health

Exclusion Criteria:

* HRT in the last 4 weeks before study entry
* treatment with non-hormonal climacteric drug (including TCM and nutritional supplement) and use of food which can interfere with menopausal symptoms during the last week before study entry or during the wash-out period before the first KMI evaluation
* treatment with drugs (including phytotherapeutics) of the ATC groups N03, N05 or N06 during the last four weeks before study entry or during the wash-out period before the first KMI evaluation
* BMI > 28 kg/m2
* thickness of uterine intima equal or more than 5 mm (only in patients with amenorrhea of 12 months or longer) or more than 15 mm (only in patients with amenorrhea of less than 12 months)
* irregular gynecological bleeding in the last 4 weeks before start of study medication without an endometrial carcinoma ruled out
* cervical smear (ASCUS) expressed anything of as follows: intraepithelial pathologic change (CIN1, CIN2, CIN3, carcinoma in situ), squamous carcinoma
* hysterectomy or supracervical hysterectomy
* more than eight years amenorrhea
* contraindication of tibolone
* cancer
* severe disease (e.g. ...) which could mask the climacteric complaints or the treatment of which could interfere with the study objectives. For example, ...
* diseases which could influence the baseline measurement of the KMI
* drug abuser, alcohol addicts, etc.
* participation in another clinical trial of phase I, II during the last 180 days or of phase III, IV during the last 90 days before study entry, or simultaneous participation in another clinical trial
* other circumstances that make the investigator expect an incomplete study participation of the patient

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240
Dates: Start 2004-09; Study Completion 2005-05

PRIMARY OUTCOMES:
Benefit-risk-balance = combination of the Mann-Whitney values (MWV) of the KMI and the frequency of adverse events at end of treatment

SECONDARY OUTCOMES:
Kupperman Menopause Index (KMI)
KMI based responder rate
CGI 1
CGI 2
CGI 3.1
subject's global assessment of efficacy
assessments of adverse events
physical examinations
global assessment of tolerability
laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Wenpai Bai, MD PhD, Principal Investigator — The First Hospital of Peking University
Locations (5):
- China (5):
  - Department of Gynecology, First Hospital of Peking University, Beijing
  - Department of Gynecology, General Hospital of PLA, Beijing
  - Department of Gynecology, Third Hospital of Peking University, Beijing
  - Department of Gynecology, West China Second Hospital of Sichuan University, Chengdu
  - Department of Gynecology, Jiangsu Province People's Hospital, Nanjing